CLINICAL TRIAL: NCT00867516
Title: A Study to Determine the Safety, Efficacy, and Pharmacokinetics of 80,160 and 320mg ALD518 Versus Placebo Administered as Multiple IV Infusions to Patients With Active Rheumatoid Arthritis Who Have Had an Inadequate Response to Methotrexate
Brief Title: Safety, Efficacy and Pharmacokinetics Study of ALD518 in Patients With Active Rheumatoid Arthritis
Acronym: ALD518-003
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALD518-CLIN-003
Record Dates: First submitted 2009-03-20; First posted 2009-03-23 (Estimated); Last update posted 2020-07-09 (Actual); Status verified 2017-09

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — clazakizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): ALD518 80 mg
  Interventions: Biological: ALD518
- 2 (Experimental): ALD518 160 mg
  Interventions: Biological: ALD518
- 3 (Experimental): ALD518 320 mg
  Interventions: Biological: ALD518
- 4 (Placebo Comparator): No ALD518
  Interventions: Biological: Infusion without ALD518'

INTERVENTIONS:
Biological: ALD518 — Two doses of ALD518, each given in an infusion of normal saline, IV over 1 hour, at Weeks 1 and 8
  Arms: 1; 2; 3
Biological: Infusion without ALD518' — 250 cc Normal saline IV over one hour Weeks 1 and 8.
  Arms: 4

SUMMARY:
The purpose of this study is to determine the safety and efficacy of ALD518 in three different doses in patients who have not had an adequate response to methotrexate.

DETAILED DESCRIPTION:
This will be a phase II, parallel-group, double-blind, randomized, placebo-controlled study of ALD518 in patients with active RA with an inadequate response to methotrexate.

Enrolled patients will be screened within a 4-week period (Day -35 to -7). within a 12-day period (Day-14 to -3) before initial dosing on Day 1 patients will be randomized to one of the following four treatment groups:

Group A: 2x ALD518 80 mg Group B: 2x ALD518 160 mg Group C: 2x ALD518 320 mg Group D: 2x placebo

In all treatment groups patients will continue to take a stable dose of methotrexate.

There will be a total of 11 visits. The total duration of the patient study participation will be approximately 16 weeks (excluding the screening period).

ELIGIBILITY:
Inclusion Criteria:

* Active Rheumatoid Arthritis for at least 16 weeks duration
* Have a C-reactive protein (CRP) of ≥ 10mg/L
* Have a stable dose of methotrexate (≥ 10mg/week) for at least 3 months

Exclusion Criteria:

* Arthritis onset prior to 16 years old
* Received any biologic therapy in the previous 12 months
* A history of or currently have active tuberculosis
* Any clinically significant concurrent medical condition

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2008-10; Primary Completion 2009-06 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of AEs and SAEs during the study | During entire length of study

SECONDARY OUTCOMES:
To evaluate the difference in treatment with ALD518 relative to treatment with placebo in the proportion of patients achieving a 20% improvement in ACR response (ACR20) at Week 12 | 12 weeks after Dose 1

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Smith, MD, FRCP, Study Director — Alder BioPharmaceuticals
Locations (26):
- Canada (2):
  - K-W Musculoskeletal Research, Inc., Kitchener, Ontario
  - Rheumatology Research Associates, Ottawa, Ontario
- Georgia (2):
  - V. Tsitlanadze Scientific Practical Centre of Rheumatology, Tbilisi
  - Medulla Chemotherapy and Immunotherapy Clinic, Tbilisi
- India (5):
  - Chanre Rheumatology and Immunology Center and Research, Malleshwaram, Bangalore
  - KLE Society Hospital and Medical Research Centre, Nehru Nagar, Belgaum
  - Sushrut Hospital, Research Centre & Post Graduate Institute of Orthopaedics, Ramadaspeth, Nagpur
  - St. John's Medical College Hospital, Bangalore
  - Krishna Institute of Medical Sciences Ltd., Secunderabad
- Poland (5):
  - Miriada Center Private Clinic of Professor Sierakowski, Bialystok
  - Nonpublic Centre of Medical Care Reumed, Lublin
  - NOVAMED - Medical Center of Poznan, Poznan
  - Provincional Rheumatological Complex named after Dr Jadwiga Titz-Kosko, Sopot
  - Szezecin Clinic of Rheumatology and Internal Diseases, Szczecin
- Russia (10):
  - Regional Clinical Hospital of War Veterans, Kemerovo
  - Institute of Clinical and Experimental Lymphology, Novosibirsk
  - Ryazan Regional Clinical Cardiologic Dispensary, Ryazan
  - Saint Petersburg Medical Academy of Postgraduate Study, Saint Petersburg
  - Saint-Petersburg State Medical Academy named after I. I. Mechnikov, Saint Petersburg
  - City Hospital #26, Saint Petersburg
  - Regional War Veterans' Hospital, Saratov
  - Tomsk Regional Clinical Hospital, Tomsk
  - Tula Regional Clinical Hospital, Tula
  - Clinical Hospital of Emergency Care named after N.V. Solovyev, Yaroslavl
- Serbia (2):
  - Institute of Rheumatology, Belgrade
  - Institute for Rehabilitation and Treatment Niska Banja, Niška Banja